CLINICAL TRIAL: NCT04610983
Title: Bioavailability of Omega-3 Long-chain Polyunsaturated Fatty Acids (LCPUFA) From Foods Enriched With Vegetable-encapsulated Omega-3 Oils
Brief Title: Omega-3 Bioavailability From Vegetable-omega-3 Enriched Products
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Commonwealth Scientific and Industrial Research Organisation, Australia (Other Government)
Collaborators: Agency for Science, Technology and Research (Other)
Responsible Party: Principal Investigator, Bradley Klingner, Project Manager and Principal Investigator delegate, Commonwealth Scientific and Industrial Research Organisation, Australia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: OBP001
Record Dates: First submitted 2020-10-26; First posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Lifestyle

STUDY DESIGN:
Intervention Model Description: A randomised, controlled, acute, 3-way cross-over study design will be used
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Experimental): Control 2 * Gel Encapsulated Algal Oil Capsules (each containing 200mg DHA) Total dose of 400mg DHA.
  Interventions: Dietary Supplement: Experimental: Control
- Treatment 1 - Semi-Solid food matrix (Experimental): Vegetable encapsulated algal oil integrated with a semi-solid food product (soup) to deliver 400 mg DHA.
  Interventions: Dietary Supplement: Experimental: Treatment 1 - Semi-Solid food matrix
- Treatment 2 - Solid food matrix (Experimental): Vegetable encapsulated algal oil integrated with a solid food product (extruded snack) to deliver 400 mg DHA.
  Interventions: Dietary Supplement: Treatment 2 - Solid food matrix

INTERVENTIONS:
Dietary Supplement: Experimental: Control — 2 x algal oil gel capsules delivering 400mg DHA in total
  Arms: Control
Dietary Supplement: Experimental: Treatment 1 - Semi-Solid food matrix — Test Food 1: 200g serve soup + "ingredient"
  Arms: Treatment 1 - Semi-Solid food matrix
Dietary Supplement: Treatment 2 - Solid food matrix — Test Food 2: 50g serve extruded snack (savoury snack) + "ingredient"
  Arms: Treatment 2 - Solid food matrix

SUMMARY:
CSIRO's Food Program has developed a novel vegetable-based Omega-3 long-chain polyunsaturated fatty acid (Omega 3)encapsulant to be used as ingredient in various food products, however, it is unknown whether the vegetable-based carrier matrix will affect omega-3 bioavailability. This project aims to compare the bioavailability of omega-3 from two test foods containing vegetable (cauliflower)-encapsulated algal oil (the "ingredient") against a control test product (algal oil gel capsules) across two ethnicities (Australian European vs. Chinese Singaporean).

DETAILED DESCRIPTION:
Omega-3 long-chain polyunsaturated fatty acids (omega-3) (eicosapentaenoic acid [EPA] and docosahexaenoic acid [DHA]) is associated with many health benefits including improved brain, heart, joint and eye health. However, <20% of the world's population consume adequate amounts of these fatty acids. Individuals who don't consume fish (major dietary omega-3 source) and particularly vegans/vegetarians are at greatest risk of omega-3 deficiency. Convenient strategies empowering consumers to increase their omega-3 intake have potential to significantly impact health outcomes. CSIRO's Food Program has developed a novel vegetable-based omega-3 encapsulant to be used as ingredient in various food products. Using algal oil as omega-3 source provides vegan/vegetarian options. However, it is unknown whether the vegetable-based carrier matrix will affect omega-3 bioavailability. As these products are intended for global markets, it is also unknown whether ethnic differences may affect omega-3 bioavailability. This project forms part of a larger project aiming to develop sensorially and culturally acceptable food products that incorporate vegetable-encapsulated omega-3 oils to assist Australian and Singaporean consumers to achieve their omega-3 LCPUFA intake. This component of the project aims to compare the bioavailability of omega-3 from two test foods containing vegetable (cauliflower)-encapsulated algal oil (the "ingredient") against a control test product (algal oil gel capsules) across two ethnicities (Australian European vs. Chinese Singaporean). To achieve this, two clinical trials, following the same protocol, will be executed in both Australia (Australian European) and Singapore (Chinese Singaporean).

ELIGIBILITY:
Inclusion Criteria:

* Healthy men
* Age: 21-50 years old
* BMI 18-27.5 kg/m2
* Consume less than 2 meals of fatty fish/week
* Not consume fish oil supplements over the past 3 months
* Identify as Australian European in ethnicity (Australian with European heritage) for Australian arm of study
* Identify as Chinese Singaporean in ethnicity (Singaporean with Chinese heritage) for Singaporean arm of study

Exclusion Criteria:

* History of chronic disease - cancer, type 2 diabetes, cardiovascular disease, liver disease or any condition that may, in the opinion of the principle investigator, influence the study outcomes (Self reported, no clinical testing will be performed)
* History of gastrointestinal disease, pancreatic insufficiency, conditions resulting in fat malabsorption - chronic pancreatitis, cystic fibrosis, coeliac disease, Crohns disease, gastric bypass surgery, small bowel resection, abnormal thyroid function (Self reported, no clinical testing will be performed)
* Bleeding disorders, currently taking anticoagulants or has received anticoagulants within 28 days of Day 1 of the trial, with the exception of low dose aspirin up to150 mg daily (Self reported)
* Any medical procedures deemed by the principal investigator to affect study outcomes
* Known food allergies, hypersensitivity, dietary avoidance or intolerance to the study foods
* Taking medications/supplements known to influence lipid metabolism and gastric emptying
* On any weight-loss program
* History of smoking during the 6 months prior to the study (Self reported)
* Persons considered by the investigator to be unwilling, unlikely or unable to comprehend or comply with the study protocol
* History of drug abuse or alcoholism (Self reported)
* Participation in another research study within 30 days preceding the start of this study

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-11-16 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Blood Plasma Omega-3 Concentration | 0 Minutes (T0), 120 Minutes (T1), 240 Minutes (T2), 360 Minutes (T3), 480 Minutes (T4) and 1440 Minutes (T5)
  Blood Plasma Omega-3 Concentration

CONTACTS AND LOCATIONS:
Locations (2):
- CSIRO, Health and Biosecurity, Adelaide, South Australia, Australia
- A*STAR, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stonehouse W, Klingner B, Tso R, Teo PS, Terefe NS, Forde CG. Bioequivalence of long-chain omega-3 polyunsaturated fatty acids from foods enriched with a novel vegetable-based omega-3 delivery system compared to gel capsules: a randomized controlled cross-over acute trial. Eur J Nutr. 2022 Jun;61(4):2129-2141. doi: 10.1007/s00394-021-02795-7. Epub 2022 Jan 18. PMID 35041046

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/83/NCT04610983/Prot_SAP_000.pdf